CLINICAL TRIAL: NCT04236349
Title: Tuberculosis Cohort in the North of Paris: Pilot Phase
Brief Title: Tuberculosis Cohort in the North of Paris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2016FM961
Record Dates: First submitted 2020-01-10; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Tuberculosis; Extra Pulmonary Tuberculosis
Keywords: Tuberculosis, cohort, lost of follow up
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Extrapulmonary; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — biological collection (DNA library; RNA library; plasma library; cell library)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CO1TB: observational: patients with pulmonary and extrapulmonary tuberculosis
- CO2TB: immunogenetics: patient with pulmonary and extrapulmonary tuberculosis and meet the following criteria:
  * informed consent form signed by the patient or by the representative of parental authority
  * affiliation to social security (beneficiary or assignee)
  * HIV negative
  Interventions: Genetic: immunogenetics

INTERVENTIONS:
Genetic: immunogenetics — blood samples at day 0, week 2, month 2; at the end of treatment (month 6 or month 9 or month 12 depend on treatment duration)
  Groups: CO2TB: immunogenetics

SUMMARY:
Tuberculosis (TB) is the leading cause of death from infectious disease in the world, just behind HIV / AIDS. Since 2005, the department of Seine Saint Denis, the poorest of France with difficult socio-economic conditions, has the highest incidence rate in metropolitan France, higher than that of Paris. In 2012, the rate of reporting was 10 times higher among people born abroad compared to those born in France, with the highest rates found among people born in sub-Saharan Africa and Asia.

It is proposed to establish for the first time in France a cohort of patients with TB disease to better understand the characteristics of patients with adverse treatment outcomes and propose solutions to achieve better control of TB. This study would recruit 200 patients per year for 5 years associated with 5 years of follow-up for a total duration of the study which would be 10 years. Given the economic stakes induced by such a study, a pilot feasibility study will be carried out initially. This smaller cohort over a shorter inclusion and follow-up period will make it possible to assess the feasibility of the large-scale cohort (princeps cohort) and to propose possible improvements to the protocol or questionnaire if problems arise in the future after achievement of this pilot study.

DETAILED DESCRIPTION:
There are flagrant shortcomings in the health care pathways of patients with TB, with a significant proportion of unknown treatment outcomes, including a large number of those lost to follow-up secondary transmission, tuberculosis recurrence, and emergence from tuberculosis. resistances. Unknown treatment outcomes are treatment outcomes not reported at 12 months of treatment initiation (lost to follow-up, transfer, no information). Health actors must mobilize to better understand the characteristics of patients with incomplete treatment outcomes and to provide solutions for better control of tuberculosis in our region. This study also want to evaluate the relationship between plasma concentrations of major antituberculosis drugs (rifampicin and isoniazid) and treatment outcomes. This study propose to constitute for the first time in France a cohort of patients presenting a TB disease in order to meet these objectives.The original study would recruit 200 patients per year for 5 years associated with 5 years of follow-up for a total duration of the study estimated at 10 years. Given the economic stakes involved in such a study, a pilot feasibility study is carry out, which is the subject of this research protocol. This smaller cohort over a shorter inclusion and follow-up period will make it possible to evaluate the feasibility of the large-scale cohort, to propose possible improvements of the protocol if problems are raised at the end of the study and launch the cohort at the same time if the study is considered feasible. A cohort should be as representative as possible of the population and the pathology studied. Thus, the population to be studied here corresponds to any adult patient or child with TB disease confirmed, consulting or hospitalized in one of the six participating services, and initiating treatment in the center. As part of the pilot study, a 1-year follow-up will be conducted to assess the feasibility of the original study. This duration is appropriate and sufficient for a first evaluation of the distribution of treatment outcomes at 1 year follow-up in the context of a study, in accordance with World Health Organisation (WHO) recommendations. Nevertheless, this one-year follow-up will only partially capture the risk of tuberculosis relapses, as part of the pilot study. This, however, will indirectly reflect the quality of the patient management system and thus assess the feasibility of the original study. It is an observational study of prospective multicentric cohort type, initially piloting, then intended to be extended by a larger original study, if it is considered feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly admitted to a consultation or hospitalization at a participating facility
* Patient with pulmonary or extrapulmonary tuberculosis confirmed on a suggestive bacteriology (direct examination, GeneXpert MTB / RIF PCR and / or culture positive) or evocative histology (evocative aspect with gigantocellular epithelioid granuloma with or without caseous necrosis) or suspicion of tuberculosis not confirmed with introduction of anti-tuberculosis treatment

Exclusion criteria :

* Refusal to give one's non-opposition to participate in the study
* Patient on antituberculous treatment for more than 21 days at the inclusion visit
* Patient already participating in another research protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with pulmonary or extrapulmonary tuberculosis
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of known treatment outcomes | 1 year

SECONDARY OUTCOMES:
number of inclusions by center | 1 year
Number of opposition to study participation among eligible patients | 1 year
Number of lost to follow-up | 1 year
Number of variables filled in for each consultation or follow-up call | At: inclusion (Day 0), Week 2 (w2), 1st month (M1), 2nd month (M2), 6th month (M6), 12th month (M12)
Genetics: identification of rare variants with strong effect for the earliest forms of pulmonary tuberculosis (before 25 y.o) and / or belonging to families with several patients and / or with recurrent forms of tuberculosis. | Day 0
  secondary outcome for CO2TB patients. rare variants with strong effect will be identified with Whole Exome sequencing method
immunology: identification of pro or anti inflammatory markers | Day 0, week 2, month 2; at the end of treatment (month 6 or month 9 or month 12 depend on treatment duration)
  secondary outcome for CO2TB patients

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenne, Bobigny, Seine Saint Denis, France